CLINICAL TRIAL: NCT02874989
Title: Targeted Removal of Pro-Inflammatory Cells: An Open Label Human Pilot Study in Idiopathic Pulmonary Fibrosis
Brief Title: Targeting Pro-Inflammatory Cells in Idiopathic Pulmonary Fibrosis: a Human Trial
Acronym: IPF
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Collaborators: Mayo Clinic (Other); The University of Texas Health Science Center at San Antonio (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: IRB00037000
Record Dates: First submitted 2016-08-17; First posted 2016-08-22 (Estimated); Last update posted 2020-05-12 (Actual); Status verified 2019-12

CONDITIONS: Idiopathic Pulmonary Fibrosis (IPF)
MeSH Terms: conditions — Idiopathic Pulmonary Fibrosis | interventions — Dasatinib; Quercetin

STUDY DESIGN:
Who Masked: Participant
Masking Description: Some patients will be randomized either to placebo or study drug and other patients will go into open label.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Dasatinib + Quercetin (Experimental)
  Interventions: Drug: Dasatinib + Quercetin
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Dasatinib + Quercetin
  Arms: Dasatinib + Quercetin
Drug: Placebo
  Arms: Placebo

SUMMARY:
The study team hypothesizes that intermittent (3 doses administered over 3 consecutive days in 3 consecutive weeks) oral administration of combination Dasatinib (100 mg/d) + Quercetin (1250 mg/d) will be safe and well tolerated in patients with IPF. Treatment with D+Q will result in reduced abundance of pro-inflammatory cells within subjects over baseline. Finally, the reduction in biomarkers of cellular pro-inflammatory state will be related to no change in functional and patient reported outcomes.

ELIGIBILITY:
Inclusion Criteria:

1. Men between ages 50 and above, at the time of signing the informed consent.
2. Post-menopausal women ages 50 and above, at the time of signing the informed consent. Note: Postmenopausal is defined as 12 months of spontaneous amenorrhea determined by self-report.
3. A clinical diagnosis of IPF and characteristic chest HRCT scan (determined by panel of pulmonary radiologists) OR biopsy showing usual interstitial pneumonia (UIP).
4. Body Mass Index (BMI) within the range 19 - 39.9 kg/ m2 (inclusive), where BMI = (weight in kg) / (height in meters)2 .
5. Subjects participating in an exercise program must be willing to maintain their current activity level for the duration of the study period.
6. Patients on stable therapy with nintedanib (Ofev) or pirfenidone (Esbriet) over the past 3 months.ORPatients not taking nintedanib (Ofev) or pirfenidone (Esbriet) may be enrolled if they have previously not tolerated one of those medications or if those medications have not yet been prescribed or used by the patient.
7. Giving signed informed consent.
8. No plans to travel over the next 6 weeks.

Exclusion Criteria:

1. More than two moderate/severe IPF exacerbations within the past year Exacerbation is defined as worsening of two or more of the following major symptoms: dyspnea, sputum volume, sputum purulence OR worsening of any one major symptom together with at least one of the following additional symptoms: sore throat, colds (nasal discharge and/or nasal congestion), fever > 37.5 ° C without any explained cause, increased cough, increase wheeze.

   A moderate exacerbation is defined as an event that is associated with a new prescription for antibiotics and/or oral steroids. A severe exacerbation is defined as an event that is associated with hospitalization or emergency room visit.
2. Any moderate/severe IPF exacerbation within the past 4 weeks.
3. History of a lung transplant.
4. Use of anti-arrhythmic medications known to cause QTc prolongation.
5. Pulmonary hypertension or cor pulmonale confirmed by echocardiography or heart catheterization.
6. Myocardial infarction, angina, hospitalization for cardiac aetiology, stroke or transient ischemic attack in the past 6 months.
7. Chronic heart failure.
8. Neurologic, musculoskeletal, or other condition that in the opinion of the study physician limits subject's ability to complete study physical assessments.
9. Uncontrolled diabetes (HbA1c > 8% and fasting glucose >200 mg/dL or the current use of insulin).
10. Subjects with values outside the specified ranges for the following Key Clinical Laboratory Tests must be excluded from the study:

    Renal function: Glomerular Filtration Rate (GFR) <30 (mL/min/1.73 m2) using formulae provided in the Study Reference Manual (SRM). Note: Subjects receiving dialysis are excluded from this study.

    ALT >2xULN and bilirubin >1.5xULN (isolated bilirubin >1.5xULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
11. Current or chronic history of liver disease, or known hepatic or biliary abnormalities (with the exception of Gilbert's syndrome or asymptomatic gallstones).
12. QTcB or QTcF > 450 msec or QTc > 480 msec in subjects with Bundle Branch Block based on a single ECG.
13. Subjects with a history of malignancy that is not in complete remission for at least 2 years or 1 year for non-melanoma skin carcinoma.
14. The subject has participated in a clinical trial and has received an investigational product within the following time period prior to participation in the current study: 30 days, 5 half-lives or twice the duration of the biological effect of the investigational product (whichever is longer).
15. History of drug or alcohol abuse within 5 years prior to randomization.
16. Use of Coumadin or other anti-platelet or anti-coagulant medication. The use of aspirin is permitted.
17. Current use of quinolone antibiotics.
18. Low CBC.
19. Cognitive Impairment (MoCA score less than 21)
20. Other medical or behavioral factors that in the judgment of the principal investigator may interfere with study participation or the ability to follow the intervention

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2016-12-16 (Actual); Primary Completion 2019-06-03 (Actual); Study Completion 2019-06-03 (Actual)

PRIMARY OUTCOMES:
Percentage of pro-inflammatory expressing cells | baseline
  A skin biopsy will be obtained at baseline and the percentage of pro-inflammatory expressing cells will be recorded
Percentage of pro-inflammatory expressing cells | 4 weeks post baseline visit biopsy/ 5 days post last dose study drug
  A skin biopsy will be obtained at 4 weeks post baseline/5 days after the last dose of study medication and the percentage of pro-inflammatory expressing cells will be recorded
Blood Pressure | screening 1 week pre baseline visit
Blood Pressure | baseline visit
Blood Pressure | 4 weeks post baseline
Weight | screening 1 week pre baseline visit
Weight | baseline visit
Weight | 4 weeks post baseline
Heart Rate | screening 1 week pre baseline visit
Heart Rate | baseline visit
Heart Rate | 4 weeks post baseline
CBC (complete blood count) | screening 1 week pre baseline visit
CBC (complete blood count) | 4 weeks post baseline
Lipid Panel | screening 1 week pre baseline visit
Lipid Panel | 4 weeks post baseline
HbA1c (glycated hemoglobin) | screening 1 week pre baseline visit
HbA1c (glycated hemoglobin) | 4 weeks post baseline
CMP (comprehensive metabolic panel) | screening 1 week pre baseline visit
CMP (comprehensive metabolic panel) | 4 weeks post baseline
Plasma hsCRP (high-sensitivity C-reactive protein) | screening 1 week pre baseline visit
Plasma hsCRP (high-sensitivity C-reactive protein) | 4 weeks post baseline
Plasma IL-6 (inflammatory biomarker) | baseline
Plasma IL-6 (inflammatory biomarker) | 4 weeks post baseline
Plasma IL-6R (inflammatory biomarker) | baseline
Plasma IL-6R (inflammatory biomarker) | 4 weeks post baseline
Plasma PASP biomarkers (inflammatory biomarkers) | baseline
Plasma PASP biomarkers (inflammatory biomarkers) | 4 weeks post baseline
p16INK4a biomarker (inflammatory biomarker) | baseline
p16INK4a biomarker (inflammatory biomarker) | 4 weeks post baseline

CONTACTS AND LOCATIONS:
Overall Officials: Stephen Kritchevsky, PhD, Principal Investigator — Wake Forest Univerisity Health Sciences
Locations (2):
- United States (2):
  - Wake Forest Baptist Health, Winston-Salem, North Carolina
  - University of Texas Health Science Center, San Antonio, Texas

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Justice JN, Nambiar AM, Tchkonia T, LeBrasseur NK, Pascual R, Hashmi SK, Prata L, Masternak MM, Kritchevsky SB, Musi N, Kirkland JL. Senolytics in idiopathic pulmonary fibrosis: Results from a first-in-human, open-label, pilot study. EBioMedicine. 2019 Feb;40:554-563. doi: 10.1016/j.ebiom.2018.12.052. Epub 2019 Jan 5. PMID 30616998

DOCUMENTS (1):
  • Informed Consent Form (2018-03-12): https://cdn.clinicaltrials.gov/large-docs/89/NCT02874989/ICF_000.pdf